CLINICAL TRIAL: NCT07121946
Title: A Phase 1, Open-label, Multicenter Study of LTZ-301 in Subjects With Relapsed/Refractory Non-Hodgkin Lymphoma
Brief Title: This is a Phase 1 Study to Evaluate the Safety of LTZ-301 in Patients With Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LTZ Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LTZ-301-001
Record Dates: First submitted 2025-08-12; First posted 2025-08-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkin Lymphoma Refractory/ Relapsed; DLBCL - Diffuse Large B Cell Lymphoma; Mantle Cell Lymphoma (MCL); Follicular Lymphoma ( FL); Marginal Zone Lymphoma (MZL)
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Subjects in this arm will participate in one (1) of eight (8) escalating defined dose level cohorts. Subjects will receive up to 54 weeks of LTZ-301 intravenously.
  Interventions: Biological: LTZ-301
- Backfill Expansion (Experimental): Subjects may be dosed at levels previously declared safe to further explore safety, tolerability, and clinical activity at particular dose levels.
  Interventions: Biological: LTZ-301
- Expansion (Experimental): A dose level will be selected to enroll additional subjects to explore safety, tolerability, and clinical activity for a selected lymphoma type.
  Interventions: Biological: LTZ-301

INTERVENTIONS:
Biological: LTZ-301 — LTZ-301 will be dosed IV, in initial 28 day cycles. First cycle dosing is every week. Second through fifth cycles are dosed every 2 weeks. Sixth cycle and beyond are 21 day cycles, and are dosed once every 3 weeks.
  Arms: Dose Escalation
Biological: LTZ-301 — LTZ-301will be dosed IV, as above
  Arms: Backfill Expansion
Biological: LTZ-301 — LTZ-301will be dosed IV, as above
  Arms: Expansion

SUMMARY:
This study is a first-in-human (FIH), Phase 1, multicenter, open-label study to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and evaluate the preliminary anti-tumor activity of LTZ-301 administered as a single agent in adult subjects with relapsed or refractory B-cell non-Hodgkin lymphoma

DETAILED DESCRIPTION:
LTZ-301 is a bispecific antibody which is a Myeloid cell engager, which targets B-cells via CD79B, and triggers phagocytosis

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Relapsed or refractory to at least 2 prior systemic treatment regimens
* At least 1 bi-dimensionally measurable lesion (≥ 1.5 cm) in longest dimension
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate bone marrow, cardiac, pulmonary, renal, and hepatic function

Exclusion Criteria:

* CLL, or Richters transformation
* Prior solid organ transplant
* Prior allogeneic stem cell transplant
* ASCT within 100 days prior to the first LTZ-301 administration
* Prior CAR-T within 60 days prior to the first LTZ-301 administration
* Current central nervous system (CNS) lymphoma
* Known history of human immunodeficiency virus (HIV) seropositivity
* Active autoimmune disease
* History of clinically significant cardiovascular disease
* symptomatic deep vein thrombosis (DVT) within 3 months of enrollment
* History of other malignancy within 3 years prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 54 weeks
  To determine the incidence of adverse events according to CTCAE v5.0 and meeting protocol defined and dose limiting toxicity criteria.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Tennessee Oncology, Nashville, Tennessee
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No